CLINICAL TRIAL: NCT02678104
Title: The Influence of Intra-alveolar Application of Honey on Healing Following Molar Teeth Extraction: A Randomized Clinical Trial
Brief Title: The Influence of Intra-alveolar Application of Honey on Healing Following Extraction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Nedal Abu-Mostafa, Dr., Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FRP/2016/23
Record Dates: First submitted 2016-01-24; First posted 2016-02-09 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Dry Socket
Keywords: Dry Socket; Honey; Tooth Extraction
MeSH Terms: conditions — Dry Socket | interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine mouth wash (Experimental): Tooth extraction. The patients will start using Chlorhexidine mouthwash on 2nd day of extraction twice daily for 7 days.
  Interventions: Procedure: Tooth extraction; Drug: Chlorhexidine mouth wash
- Manuka Honey (Experimental): intra-alveolar application of Manuka Honey after tooth extraction.
  Interventions: Procedure: Tooth extraction; Drug: Intra-alveolar application of Manuka Honey

INTERVENTIONS:
Procedure: Tooth extraction — Tooth removal
Drug: Chlorhexidine mouth wash — Chlorhexidine mouth wash
  Other Names: Oraxine 0.2% Chlorhexidine mouth wash
  Arms: Chlorhexidine mouth wash
Drug: Intra-alveolar application of Manuka Honey — Intra-alveolar application of Manuka Honey directly after extraction.
  Other Names: Marks & Spencer Manuka Honey
  Arms: Manuka Honey

SUMMARY:
A prospective randomized parallel trial will be carried out on 100 patients who have extraction of single molar tooth. Teeth extractions will be done under local anesthesia. The patients will be divided randomly into two parallel groups. Group 1: The patients will start using Chlorhexidine mouthwash on the second day of extraction twice daily for 7 days. Group 2: After extraction, Manuka Honey will be applied topically into the extraction socket. Postoperative instructions will be given for all patients in addition to the prescription of ibuprofen 600 mg every 8 hours for 3 days.

Re-evaluation:

Postoperative day 3: tenderness with probing the socket, empty socket, food debris, halitosis and assessment of pain. For group 2, the intra-alveolar application of honey will be repeated. Re-evaluation will be repeated in the seventh post-operative day. Acute alveolar osteitis, (dry socket) is diagnosed if the patient presented between the 2nd and 4th days with pain or tenderness in the socket with probing, empty socket and food debris with or without halitosis.

DETAILED DESCRIPTION:
A prospective randomized experimental parallel trial will be carried out on 100 male and female patients who have extraction of single molar tooth. Extractions will be performed by dental interns or dental students under supervision of surgery instructors in the Colleges' Clinics.

The study has been registered in the College's Research Center, with a registration number of FRP/2016/23. It will follow the World Medical Association Declaration of Helsinki, the patients will be informed about the objectives of the study, and informed consent has to be signed. All required information was documented in the questionnaire paper regarding name, age, gender, mobile number, file number, smoking, medical condition, tooth indicated for extraction, pre-operative pain and halitosis.

Teeth extractions will be done under local anesthesia. Simple extractions will be done by elevators and forceps, while root separations will be done using a surgical handpiece and burs with normal saline irrigation.

The patients will be divided randomly into two parallel groups by asking them to choose 1 out of 100 playing cards. These cards, which have images of different shapes, have been mixed. The first shape includes 50 cards and represents the first study group, while the second shape includes 50 cards and represents the second study group.

Both groups will receive a bottle of 0.2 % Chlorhexidine mouthwash. Group 1: The patients will start using Chlorhexidine mouthwash on the second day of extraction twice daily for 7 days. Group 2: After tooth extraction, Manuka Honey will be applied topically by a cotton swab into the extraction socket.

Follow up:

The patients will be followed in the third postoperative day. Re-evaluation includes tenderness with probing the socket, empty socket, and assessment of pain by (VAS) from (0, 1, 2,….10). Score 0 representing no pain, 10 representing severe pain. Re-evaluation will be repeated in the seventh post-operative day including the same evaluation points of the third day.

Acute alveolar osteitis, (dry socket) is diagnosed if the patient presented between the 2nd and 4th days with pain or tenderness in the socket with probing, empty socket.

Frequencies and percentages are calculated for qualitative data (SPSS software version.22). Chi-square test will be applied to compare both subgroups.

ELIGIBILITY:
Inclusion criteria:

* Patients who have extraction of single molar tooth

Exclusion criteria:

* Patients with uncontrolled systemic diseases
* Pregnant women
* Breastfeeding women
* Women are using oral contraceptives
* Allergy to chlorhexidine
* Allergy to honey
* Presence of acute infection, cystic lesions
* Traumatic extraction
* Extraction requiring bone reduction
* Extractions lasted more than 30 minutes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pain day 3 | on the 3rd day
  Assessment of pain by (VAS) from (0, 1, 2,….10).

SECONDARY OUTCOMES:
Empty socket day 3 | on the 3rd day
  By inspection. The socket is empty and does not contain blood clot
Empty socket day 7 | in the 7th day
  By inspection. The socket is empty and does not contain blood clot
Tenderness within the socket day 3 | on the 3rd day
  By probing the socket
Tenderness within the socket day 7 | on the 7th day
  By probing the socket
Pain day 7 | on the 7th day
  Assessment of pain by (VAS) from (0, 1, 2,….10).

CONTACTS AND LOCATIONS:
Overall Officials: Nedal A Abu Mostafa, Lecturer, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- RiyadH Colleges of dentistry and Pharmacy, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu-Mostafa NA, Alqahtani A, Abu-Hasna M, Alhokail A, Aladsani A. A randomized clinical trial compared the effect of intra-alveolar 0.2 % Chlorohexidine bio-adhesive gel versus 0.12% Chlorohexidine rinse in reducing alveolar osteitis following molar teeth extractions. Med Oral Patol Oral Cir Bucal. 2015 Jan 1;20(1):e82-7. doi: 10.4317/medoral.19932. PMID 25475768
- [Background] Alexander RE. Dental extraction wound management: a case against medicating postextraction sockets. J Oral Maxillofac Surg. 2000 May;58(5):538-51. doi: 10.1016/s0278-2391(00)90017-x. No abstract available. PMID 10800910
- [Background] Bloomer CR. Alveolar osteitis prevention by immediate placement of medicated packing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2000 Sep;90(3):282-4. doi: 10.1067/moe.2000.108919. PMID 10982947
- [Background] Caso A, Hung LK, Beirne OR. Prevention of alveolar osteitis with chlorhexidine: a meta-analytic review. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Feb;99(2):155-9. doi: 10.1016/j.tripleo.2004.05.009. PMID 15660084
- [Background] Efem SE. Clinical observations on the wound healing properties of honey. Br J Surg. 1988 Jul;75(7):679-81. doi: 10.1002/bjs.1800750718. PMID 3416123
- [Background] Jull AB, Cullum N, Dumville JC, Westby MJ, Deshpande S, Walker N. Honey as a topical treatment for wounds. Cochrane Database Syst Rev. 2015 Mar 6;2015(3):CD005083. doi: 10.1002/14651858.CD005083.pub4. PMID 25742878
- [Background] Nasir NA, Halim AS, Singh KK, Dorai AA, Haneef MN. Antibacterial properties of tualang honey and its effect in burn wound management: a comparative study. BMC Complement Altern Med. 2010 Jun 24;10:31. doi: 10.1186/1472-6882-10-31. PMID 20576085
- [Background] Pieper B. Honey-based dressings and wound care: an option for care in the United States. J Wound Ostomy Continence Nurs. 2009 Jan-Feb;36(1):60-6; quiz 67-8. doi: 10.1097/01.WON.0000345177.58740.7d. PMID 19155824
- [Background] Singh V, Pal US, Singh R, Soni N. Honey a sweet approach to alveolar osteitis: A study. Natl J Maxillofac Surg. 2014 Jan;5(1):31-4. doi: 10.4103/0975-5950.140166. PMID 25298714
- [Result] Atwa AD, AbuShahba RY, Mostafa M, Hashem MI. Effect of honey in preventing gingivitis and dental caries in patients undergoing orthodontic treatment. Saudi Dent J. 2014 Jul;26(3):108-14. doi: 10.1016/j.sdentj.2014.03.001. Epub 2014 Apr 19. PMID 25057231